CLINICAL TRIAL: NCT04392245
Title: A Worldwide Survey on Proctologic Practice During Covid-19 Lockdown
Brief Title: Proctologic Practice and Covid-19
Acronym: PROCTOLOCK
Status: Completed | Type: Observational
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Collaborators: Gaetano Gallo (Unknown); Alessandro Sturiale (Unknown); Veronica De Simone (Unknown); Gian Luca Di Tanna (Unknown); Iacopo Giani (Unknown); Ugo Grossi (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Proctologic Practice During COVID-19
Keywords: proctology; covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross-sectional non-incentivized worldwide web survey.

A worldwide survey of 1050 respondents showed that proctologic practice has been seriously affected by the pandemic. Age, gender and level of hospital preparedness predicted the change of status of surgical and outpatient activities.

The results of our study may inform the development of strategies to reopen activities while protecting frontline healthcare workers.

DETAILED DESCRIPTION:
A 27-item survey (namely, 'ProctoLock 2020') was designed and developed by the authors using an online platform ('Online surveys' [formerly BOS - Bristol Online Survey], developed by the University of Bristol) in accordance with the American Association for Public Opinion Research (AAPOR) guidelines and the Checklist for Reporting Results of Internet E-Surveys [CHERRIES]

ELIGIBILITY:
Inclusion Criteria:

Members of renowned scientific societies with an interest in coloproctology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Experts in the field who joined a previous qualitative study[15] (N=492) were invited to complete a web survey (participants could be identified only via their valid email address; no other identifying information was collected). The survey link was sent to scientific societies of interest to coloproctologists (i.e. Italian Society of Colorectal Surgery, Russian Association of Coloproctologists, Mediterranean Society of Coloproctology) and disseminated to their members. All collaborators (ProctoLock 2020 Working Group) committed to further recruitment of participants by direct invitation. Participation was entirely voluntary with no compensation offered. Informed consent was obtained from all those agreeing to complete a survey. This study was exempt from review board approval at authors' institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Predictive power of respondents' and hospitals' demographics on the change of status of proctologic surgical and outpatient activities | April 15th to 26th 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Gallo Gallo, Catanzaro, Italy

REFERENCES:
- [Derived] Gallo G, Sturiale A, De Simone V, Mancini S, Di Tanna GL, Milito G, Bianco F, Perinotti R, Giani I, Grossi U; ProctoLock2020 Working Group; Aiello D, Bianco F, Bondurri A, Gallo G, La Torre M, Milito G, Perinotti R, Pietroletti R, Serventi A, Fiorino M, De Simone V, Grossi U, Manigrasso M, Sturiale A, Zaffaroni G, Boffi F, Bellato V, Cantarella F, Deidda S, Marino F, Martellucci J, Milone M, Picciariello A, Bravo AM, Vigorita V, Cunha MF, Leventoglu S, Garmanova T, Tsarkov P, El-Hussuna A, Frontali A, Ioannidis A, Bislenghi G, Shalaby M, Porzio FC, Wu J, Zimmerman D, Elbetti C, Mayol J, Naldini G, Trompetto M, Sammarco G, Santoro GA. Deadlock of proctologic practice in Italy during COVID-19 pandemic: a national report from ProctoLock2020. Updates Surg. 2020 Dec;72(4):1255-1261. doi: 10.1007/s13304-020-00860-0. Epub 2020 Aug 8. PMID 32770466